CLINICAL TRIAL: NCT03815643
Title: An Open-Label, Multicenter Follow-up Study to Collect Long-term Data on Participants From Multiple Avelumab (MSB0010718C) Clinical Studies
Brief Title: Avelumab Program Rollover Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS100070_0176; 2018-003711-21 (EudraCT Number); 2024-514274-46-00 (EU CTIS Number)
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumors
Keywords: Avelumab; Non-small cell lung cancer (NSCLC); Renal cell carcinoma (RCC); Urothelial carcinoma (UC); Ovarian cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Ovarian Neoplasms | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab (Experimental)
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Participants entering this roll over study will receive avelumab as a 1-hour intravenous (IV) infusion at 10 milligram per kilogram (mg/kg) once every 2 weeks until progressive disease, according to respective parent studies (EMR100070-001, EMR100070-002, EMR100070-004 and EMR100070-008).
  Other Names: MSB0010718C

SUMMARY:
The main purpose of this study is to monitor the safety and tolerability of avelumab in participants with solid tumors who continue treatment with avelumab under the same treatment regimen as in the parent avelumab study.

ELIGIBILITY:
Inclusion Criteria:

* Participants under enrollment and treatment in an avelumab clinical study under the sponsorship of EMD Serono Research & Development Institute, Inc. / Merck KGaA, Darmstadt, Germany

  * Merck Serono Co., Ltd (Japan)
* Participants currently enrolled in an avelumab parent study and are on active treatment with avelumab or in long-term survival follow-up after treatment
* Participants on active treatment must agree to continue to use highly effective contraception (that is, methods with a failure rate of less than 1% per year) for both male and female participants if the risk of conception exists
* Other protocol defined inclusion criteria could apply.

Exclusion Criteria:

* Participants who are pregnant or breastfeeding
* Participants still on active treatment: Known hypersensitivity to any of the study intervention ingredients
* Participant has been enrolled in the comparator arm of avelumab parent study
* Participant has been withdrawn from avelumab parent study for any reason
* Any other reason that, in the opinion of the Investigator, precludes the participant from participating in the study
* Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2027-02-19 (Estimated); Study Completion 2027-02-19 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Treatment-related Non-serious Treatment-Emergent Adverse Events (TEAEs), All Serious AEs, Immunerelated AEs and Infusion-related Reactions According to Version of National Cancer Institute Common Technology Criteria for Adverse Events | From enrollment to end of survival follow-up (up to 5 years after the last participant receives the last dose of avelumab)

SECONDARY OUTCOMES:
Overall Survival (OS) | From baseline up to 5 years
Progression Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | From baseline up to 5 years
Duration of Response (DOR) Assessed From Complete Response (CR) or Partial Response (PR) | From baseline up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (104):
- United States (26):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of California Davis Health System - Comprehensive Cancer Center, Sacramento, California
  - Providence Medical Foundation, Santa Rosa, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Norwalk Hospital - The Whittingham Cancer Center, Norwalk, Connecticut
  - Hematology - Oncology Associates of the Treasure Coast - Hematology-Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - Michigan State University, Lansing, Michigan
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Kansas City Research Institute, LLC - Phase I Unit, Kansas City, Missouri
  - University of Cincinnati - PARENT, Cincinnati, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - Oncology/Hematology Care Clinical Trials, LLC, Cincinnati, Ohio
  - OSU - James Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Greenville Hospital System University Medical Center (ITOR) - Upstate Affiliate Organization, Greenville, South Carolina
  - The West Clinic, Germantown, Tennessee
  - SCRI - Tennessee Oncology, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - Henry Ford Hospital, San Antonio, Texas
  - University of Vermont Medical Center - Fletcher Allen Gastroenterology, Burlington, Vermont
- Argentina (2):
  - Instituto Alexander Fleming, Ciudad Autonoma Buenos Aires
  - Clínica Universitaria Privada Reina Fabiola, Córdoba
- Australia (2):
  - Ballarat Health Services, Ballarat
  - Monash Medical Centre Clayton, Clayton
- Belgium (2):
  - Centre Hospitalier de l'Ardenne - Pharmacie, Libramont
  - Clinique CHC MontLégia, Liège
- Hospital de Câncer de Barretos - Fundação Pio XII, Barretos, Brazil
- MHAT for women's health - Nadezhda, OOD, Sofia, Bulgaria
- Czechia (2):
  - Nemocnice Rudolfa a Stefanie Benesov a.s. nemocnice Stredoceskeho kraje - parent, Benešov
  - Masarykuv onkologicky ustav - 300176866 Parent, Brno
- France (11):
  - CHU Besançon - Hôpital Jean Minjoz - Service d'oncologie Medicale, Besançon
  - Centre Oscar Lambret - Service d'Oncologie medicale, Lille
  - ICO - Site Paul Papin - service d'oncologie medicale, Nantes
  - ICO - Site René Gauducheau - Service d'Oncologie medicale, Nantes
  - Centre Antoine Lacassagne - Service d'Hématologie Oncologie, Nice
  - Institut Curie - site de Paris - Service d'Oncologie Médicale, Paris
  - CHU Bordeaux - Service d'Oncologie Médicale, Pessac
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque - Unité d'Explorations Fonctionnelles Respiratoires, Pessac
  - CHU Poitiers - Hôpital la Milétrie - service d'oncologie médicale, Poitiers
  - Centre Paul Strauss - Service de Médecine Oncologique, Strasbourg
  - Hopital Larrey - Service de Pneumologie et Oncologie Thoracique, Toulouse
- Universitaetsklinikum Essen - Westdeutsches Tumorzentrum, Essen, Germany
- Hungary (2):
  - Petz Aladar Egyetemi Oktato Korhaz - Pulmonologiai Osztaly, Győr
  - Zala Varmegyei Szent Rafael Korhaz - Pulmonologiai Osztaly, Zalaegerszeg
- Italy (5):
  - Azienda Ospedaliera Universitaria- Università degli Studi della Campania "Luigi Vanvitelli" - Dipartimento Oncologia, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Oncologia Medica, Roma
  - Istituto Nazionale Tumori Regina Elena IRCCS - UOC Oncologia Medica A, Roma
  - Istituto Clinico Humanitas - U.O. di Oncologia Medica ed Ematologia, Rozzano
- Japan (8):
  - National Cancer Center Hospital (NCCH), Chūōku
  - National Cancer Center Hospital - Dept of Gastrointestinal Oncology, Chūōku
  - Osaka Habikino Medical Center - Dept of Pulmonary Oncology, Habikino-shi
  - Cancer Institute Hospital of JFCR - Dept of Respiratory Medicine, Kōtoku
  - Kurume University Hospital - Dept of Lung Cancer Center, Kurume-shi
  - Osaka City General Hospital - Dept of Clinical Oncology, Osaka
  - Tohoku University Hospital, Sendai
  - Osaka University Hospital - Dept of Gastrointestinal Surgery, Suita-shi
- Health Pharma Professional Research S.A. de C.V., México, Mexico
- Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy - Dept of Lungs and Chest Oncology, Warsaw, Poland
- Romania (5):
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta" Cluj Napoca - Sectia Radioterapie III, Cluj-Napoca
  - S.C Radiotherapy Center Cluj S.R.L - Parent, Comuna Floresti
  - Institutul Regional de Oncologie Iasi - Sectia Oncologie Medicala, Iași
  - Spitalul Clinic Municipal "Dr. Gavril Curteanu" Oradea - Centrul Oncologie Medicala, Oradea
  - S.C Oncomed S.R.L - Specialitatea Oncologie Medicala, Timișoara
- Russia (6):
  - RBIH "Kursk regional clinical oncology dispensary" of Kursk Region Healthcare Committee, Kursk
  - SBHI of Novosibirsk region "Novosibirsk Regional Oncological Dispensary", Novosibirsk
  - BHI of Omsk region "Clinical Oncology Dispensary" - Building #2, Omsk
  - FSBI "National Medical Research Center for Oncology n.a. N.N. Petrov" of the MoH of the RF - Parent, Saint Petersburg
  - LLC "Medical Technologies" - Parent, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University - PARENT, Saint Petersburg
- South Korea (9):
  - Chungbuk National University Hospital, Cheongju-si
  - Chonnam National University Hwasun Hospital, Daejeon
  - National Cancer Center, Goyang
  - Gachon University Gil Medical Center, Incheon
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau - Dept of Oncology, Barcelona
  - Hospital Universitari Vall d'Hebron - Oncology Dept., Barcelona
  - Hospital General Universitario Gregorio Marañon - Servicio de Oncologia Medica, Madrid
  - Hospital de Mataro - Servicio de Oncologia Medica, Mataró
- Songklanagarind Hospital - Department of Medicine, Songkhla, Thailand
- Turkey (Türkiye) (8):
  - Adana City Hospital - Parent Account, Adana
  - Ankara University Medical Faculty - Medical Oncology, Ankara
  - Hacettepe University Medical Faculty - Oncology, Ankara
  - Goztepe Prof. Dr. Suleyman Yalcin City Hospital - Medical Oncology, Istanbul
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty - Medical Oncology, Istanbul
  - Medipol University Medical Faculty - Parent, Istanbul
  - Ege University Medical Faculty - PARENT, Izmir
  - Mersin University Medical Faculty - Medical Oncology, Mersin
- Ukraine (3):
  - CNE KHERSON REG ONCOLOGICAL DISPENSARY OF KHERSON RC - Day Hosp of Polycl with Outpatient Chemoth Room, Kherson
  - BP Medical, Vinnytsia
  - Podilskyi Regional Oncological Center - Dept of Chemotherapy, Vinnytsia
- United Kingdom (3):
  - Sarah Cannon Research Institute UK, London
  - Mount Vernon Cancer Centre, Northwood
  - Derriford Hospital - Dept of Oncology Clinical Trials, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS100070_0176
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html